CLINICAL TRIAL: NCT00806533
Title: Infusion of Venofundin 6% or Tetraspan 6% in Paediatric Patients Aged up to 12 Years
Brief Title: Non-Interventional (Observational) Post-Authorization Safety Study of HES 130/0.42 in Paediatric Patients
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Dr. Elke von Kleist, B. Braun Melsungen AG
Other Study IDs: HC-O-H-0509
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HES 130 / 0.42: paediatric patients aged up to 12 years requiring non-emergency volume replacement therapy with HES 130/0.42
  Interventions: Drug: HES 130 / 0.42 (Venofundin 6%, Tetraspan 6%)

INTERVENTIONS:
Drug: HES 130 / 0.42 (Venofundin 6%, Tetraspan 6%) — solution for intravenous infusion applied according to SmPC
  Other Names: Venofundin 6%, Tetraspan 6%

SUMMARY:
This observational (non-interventional) post-authorization safety study (PASS) will investigate the application of Venofundin 6% and of Tetraspan 6% in children with special regard to drug safety.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤12 years
* Risk of anaesthesia: American Society of Anaesthesiologists (ASA) risk score: I - III
* infusion of Venofundin 6% or of Tetraspan 6%
* elective intervention

Exclusion Criteria:

* contraindications according to SmPC

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: paediatric patients aged up to 12 years
Sampling Method: Probability Sample
Enrollment: 1130 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
incidence of adverse events | peri-operative

CONTACTS AND LOCATIONS:
Overall Officials: R. Suempelmann, Prof. Dr., Principal Investigator — MHH Hannover
Locations (10):
- Donauspital SMZ-OST, Vienna, Austria
- Czechia (2):
  - Clinic of Children's Anaesthesiology and Resuscitation, Brno
  - Clinic of Anaesthesiology and Resuscitation, Prague
- Germany (4):
  - Klinik für Anästhesiologie und Intensivmedizin, TU Universität Dresden, Dresden
  - Klinik für Anästhesiologie und Intensivmedizin, Medizinische Hochschule Hannover, Hanover
  - Klinikum Mannheim, Mannheim
  - Olgahospital, Stuttgart
- S. Orsola Hospital, University hospital, Bologna, Italy
- Netherlands (2):
  - Academic Mesich Centrum (AMC), Amsterdam
  - Erasmus MC, Univesity Medical Center Rotterdam, Sophias's Children's Hospital (SKZ), Rotterdam

REFERENCES:
- [Background] Sumpelmann R, Kretz FJ, Gabler R, Luntzer R, Baroncini S, Osterkorn D, Haeger MC, Osthaus WA. Hydroxyethyl starch 130/0.42/6:1 for perioperative plasma volume replacement in children: preliminary results of a European Prospective Multicenter Observational Postauthorization Safety Study (PASS). Paediatr Anaesth. 2008 Oct;18(10):929-33. doi: 10.1111/j.1460-9592.2008.02696.x. Epub 2008 Jul 21. PMID 18647272